CLINICAL TRIAL: NCT02323958
Title: Effect of Transcutaneous Electrical Acupoint Stimulation on Outcome During Emergence From Anesthesia in Patients Undergoing Robotic Laparoscopic Gynecologic Surgery
Brief Title: TEAS to Improve Outcome During Emergence From General Anesthesia After Robotic Surgery
Acronym: TIGER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, Dr, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XJH-A-2014-6-26-01
Record Dates: First submitted 2014-12-08; First posted 2014-12-24 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Anesthesia
MeSH Terms: interventions — Electrodes; Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Acupoint stimulation (Experimental): Electrical stimulation is given through electrodes attached to acupoints
  Interventions: Other: acupoint stimulation; Other: electrode attached; Device: electrical stimulation
- Non-acupoint stimulation (Placebo Comparator): Electrical stimulation is given through electrodes attached to non-acupoints
  Interventions: Other: non-acupoint stimulation; Other: electrode attached; Device: electrical stimulation
- Control stimulation (Sham Comparator): Electrode attached but no stimulation is given
  Interventions: Other: electrode attached

INTERVENTIONS:
Other: acupoint stimulation — stimulation is given at acupoints
  Arms: Acupoint stimulation
Other: non-acupoint stimulation — stimulation is given at acupoints
  Arms: Non-acupoint stimulation
Other: electrode attached — electrodes are attached to skin
  Other Names: electrode
Device: electrical stimulation — electrical stimulation is given through electrodes attached to th skin
  Arms: Acupoint stimulation; Non-acupoint stimulation

SUMMARY:
This study is to observe whether transcutaneous electrical stimulation at specific acupoints could improve the quality of emergence in patients undergoing robotic laparoscopic gynecologic surgery.

DETAILED DESCRIPTION:
During robotic laparoscopic gynecologic surgery, the patients are put in an extremely trendelenburg positon. And a long duration of this position could lead to delayed emergence or agitation. Stimulation at some acupoints were reported to improve homeostasis. In this study we tend to observe whether transcutaneous electrical stimulation at specific acupoints could improve the quality of emergence in patients undergoing robotic laparoscopic gynecologic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for robotic laparoscopic gynecologic surgery under general anesthesia
* Patients with written informed consent

Exclusion Criteria:

* Patients with difficulty in communication
* Patients with disease of central nervous system

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-12; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Time to awake | from end of inhaling sevoflurane to departing from postanesthesia care unit(PACU),an anticipated average of 1 hour
  time to open eyes to verbal command

SECONDARY OUTCOMES:
Richmond Score | from end of inhaling sevoflurane to departing from PACU,an anticipated average of 1 hour
  status of the patients during emergence
Time to extubation | from end of inhaling sevoflurane to departing from PACU,an anticipated average of 1 hour
QoR-15 | from end of inhaling sevoflurane to 24h after surgery,an anticipated average of 24 hour
  Score of quality of recovery using a 15 items questionaire
residual sedation | from arriving at PACU to departing from PACU,an anticipated average of 30min
PONV | from arriving at PACU to departing from PACU,an anticipated average of 30min
  postoperative nausea and vomiting in the PACU
VAS score | from arriving at PACU to departing from PACU,an anticipated average of 30min
  visual analogue score of pain in the PACU, scored 0-10
serum Aquaporin 4 | from before anesthesia to after surgery, an anticipated average of 4 hours
  level of serum Aquaporin 4 before anesthesia and at the end of the surgery
serum MMP9 | from before anesthesia to after surgery, an anticipated average of 4 hours
  level of serum Matrix metallop roteinase before anesthesia and at the end of the surgery
serum S100β | from before anesthesia to after surgery, an anticipated average of 4 hours
  level of serum S100β before anesthesia and at the end of the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hailong Dong, PhD, Study Chair — Air Force Military Medical University, China
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Result] Schramm P, Treiber AH, Berres M, Pestel G, Engelhard K, Werner C, Closhen D. Time course of cerebrovascular autoregulation during extreme Trendelenburg position for robotic-assisted prostatic surgery. Anaesthesia. 2014 Jan;69(1):58-63. doi: 10.1111/anae.12477. Epub 2013 Nov 20. PMID 24256501
- [Result] Pandey R, Garg R, Darlong V, Punj J, Chandralekha, Kumar A. Unpredicted neurological complications after robotic laparoscopic radical cystectomy and ileal conduit formation in steep trendelenburg position: two case reports. Acta Anaesthesiol Belg. 2010;61(3):163-6. PMID 21268573